CLINICAL TRIAL: NCT00676897
Title: Study of Statin Therapy in the Treatment of Sepsis
Brief Title: Statin Therapy in the Treatment of Sepsis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Michael Donnino, Dr. Michael Donnino, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2007P000257
Record Dates: First submitted 2008-05-09; First posted 2008-05-13 (Estimated); Results first posted 2017-06-14 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-05

CONDITIONS: Septic Shock
Keywords: statin, sepsis, septic shock, simvastatin
MeSH Terms: conditions — Shock, Septic; Sepsis | interventions — Simvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Simvastatin 40 mg PO or NGT
  Interventions: Drug: Simvastatin
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Simvastatin — Simvastatin 40mg PO or NGT
  Other Names: Zocor
  Arms: 1
Drug: Placebo — Corn Starch
  Arms: 2

SUMMARY:
Simvastatin will attenutat IL-6 levels and lead to a more rapid shock reversal than placebo

ELIGIBILITY:
Inclusion Criteria:

* Greater than 18 years old
* Hypotensive requiring vasopressors
* Suspected Infection

Exclusion Criteria:

* Pregnant
* Liver Failure (ALT or AST > 120)
* Rhabomyolysis (CPK > 3x normal)
* Comfort care measures status
* Chronic Liver Disease (Cirrhosis)
* Use of Cyclosporin, Digoxin, Statins
* Patients who are unable to take medications by mouth or NGT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2008-02; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael W Donnino, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Ghosh CC, Thamm K, Berghelli AV, Schrimpf C, Maski MR, Abid T, Milam KE, Rajakumar A, Santel A, Kielstein JT, Ahmed A, Thickett D, Wang K, Chase M, Donnino MW, Aird WC, Haller H, David S, Parikh SM. Drug Repurposing Screen Identifies Foxo1-Dependent Angiopoietin-2 Regulation in Sepsis. Crit Care Med. 2015 Jul;43(7):e230-40. doi: 10.1097/CCM.0000000000000993. PMID 25855898
- [Derived] Dobesh PP, Olsen KM. Statins role in the prevention and treatment of sepsis. Pharmacol Res. 2014 Oct;88:31-40. doi: 10.1016/j.phrs.2014.04.010. Epub 2014 May 2. PMID 24794878
- [Derived] Donnino MW, Cocchi MN, Salciccioli JD, Kim D, Naini AB, Buettner C, Akuthota P. Coenzyme Q10 levels are low and may be associated with the inflammatory cascade in septic shock. Crit Care. 2011 Aug 9;15(4):R189. doi: 10.1186/cc10343. PMID 21827677

RESULTS

PARTICIPANT FLOW:
Groups:
- Statin Group: Simvastatin: Simvastatin 40mg PO or NGT
- Placebo Group: Placebo: Corn Starch
Period: Overall Study
Arm/Group | Statin Group | Placebo Group
Started | 8 | 10
Completed | 8 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Statin Group | Placebo Group | Total
Number analyzed (Participants) | 8 | 10 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (18) | 54 (16) | 58.72 (17.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 4 | 7 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 8 | 10 | 18
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 3 | 4
  White | 7 | 7 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 10 | 18

OUTCOME MEASURES:

1. Primary Outcome: Time to Shock Reversal
Time Frame: up to 7 days
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Statin Group | Placebo Group
Number analyzed (Participants) | 8 | 10
hours | 44.4 (57.3) | 28.6 (34.5)

2. Secondary Outcome: Inflammatory Marker Levels
Description: Change in inflammatory marker levels over time from time zero to time 24 hour.
Time Frame: over 24 hours (time zero and time 24 hours)
Measure: Mean (Standard Deviation); unit: pg/mL and ng/mL
Arm/Group | Statin Group | Placebo Group
Number analyzed (Participants) | 8 | 10
pg/mL and ng/mL
  VEGF (pg/mL) | -98 (306) | 269 (396)
  IL-6 (pg/mL) | -370 (698) | -423 (620)
  TNF-alpha (pg/mL) | -0.52 (26) | -2.17 (43)
  ICAM (ng/mL) | 148 (282) | -0.10 (69)
  VCAM (ng/mL) | 1279 (2275) | 190 (1049)
  eSelectin (ng/mL) | 98 (202) | 11 (29)

ADVERSE EVENTS:
Arm/Group | Statin Group | Placebo Group
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/10
Other Adverse Events (participants affected / at risk) | 0/8 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No